CLINICAL TRIAL: NCT02506023
Title: Characterization of Laboratory Response to DDAVP in Adult Hemophilia A Carriers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Robert Sidonio, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00080329
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Hemophilia A
Keywords: Factor VIII antigen; von Willebrand factor (vWF) antigen; Mutation type
MeSH Terms: conditions — Hemophilia A | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hemophilia A carriers with mild mutation (Active Comparator): Hemophilia A carriers with a mild type mutation will be given a single intravenous dose of 0.3mcg/kg of DDAVP (Desmopressin).
  Interventions: Drug: Desmopressin
- Hemophilia A Carriers with severe mutation (Active Comparator): Hemophilia A carriers with a severe type mutation will be given a single intravenous dose of 0.3mcg/kg of DDAVP (Desmopressin).
  Interventions: Drug: Desmopressin
- Control (Active Comparator): Subjects with a mild qualitative platelet dysfunction will be given a single intravenous dose of 0.3mcg/kg of DDAVP (Desmopressin).
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Desmopressin or DDAVP will be administered intravenously (IV) via a nontraumatic peripheral IV line at a dose of 0.3 mcg/kg over 30 minutes.
  Other Names: DDAVP

SUMMARY:
The purpose of this study is to determine how female hemophilia A carriers respond to a medication called DDAVP (Desmopressin).

DETAILED DESCRIPTION:
DDAVP (Desmopressin) is commonly used in the treatment of persons with bleeding disorders such as hemophilia, von Willebrand disease, or qualitative platelet disorders to help them clot better. The investigator wants to assess the increase in the subjects' clotting factors in response to intravenous DDAVP (Desmopressin) and the levels of these internal clotting factors will be measured at different times after the medication is given. The investigator will compare the response to DDAVP (Desmopressin) in adult hemophilia A carriers to women with a diagnosis of qualitative platelet dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for hemophilia A carriers:

* Females 18-60 years of age at time of enrollment
* Genetically verified or obligate hemophilia A carrier (mother of 2 boys with hemophilia A, daughter of a father with hemophilia A or mother of a son and another male relative with hemophilia A)
* To stratify patients by carriage of mutation type 10 hemophilia carriers of mild mutations that are predicted to lead to reduced FVIII secretion, protein stability or thrombin cleavage site interference and 10 hemophilia carriers of severe mutations that lead to predicted negative cross reactive material will be selected. Predicted FVIII function of the mutation will be verified by EAHAD (European Association for Haemophilia and Allied Disorders) Coagulant Factor Variant Database at www.eahad-db.org)
* Weight >40kg to ensure volumes of blood to be drawn are within accepted safe range

Inclusion criteria for non-hemophilia A carriers (Females with mild qualitative platelet dysfunction):

* Females 18-60 years of age at time of enrollment
* Whole blood or platelet rich plasma lumiaggregometry consistent with reduced aggregation to at least 1 agonist on at least one occasion (excluding evidence of Glanzmanns Thrombasthenia or Bernard Soulier Syndrome) or determined by primary hematologist as having a qualitative platelet disorder
* Age-matched by 10 years to carrier enrolled
* Weight >40kg to ensure volumes of blood to be drawn are within accepted safe range

Exclusion Criteria:

* Personal history of concomitant bleeding or clotting disorder
* Cardiac condition that requires the daily use of Aspirin or Clopidogrel
* Inability to comply with fluid restriction protocol for 24 hours following Desmopressin (DDAVP)
* Personal history of a myocardial infarction, renal or hepatic insufficiency or epilepsy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07; Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects that achieve and sustain >50% increase in Factor VIII antigen levels | 240 minutes
  After administration of intravenous Desmopressin (DDAVP) at 0.3mcg/kg, the percentage of subjects that achieve and sustain Factor VIII antigen (FVIII:C) levels >50% at 240 minutes as compared to baseline will be recorded. The levels of Factor VIII antigen (FVIII:C) will be measured using a one-stage assay. The laboratory response between carriers and the control group will be compared and the percentage of subjects that have greater than a 2-fold response from baseline and sustainment of Factor VIII antigen (FVIII:C) >50% at 240 minutes will be recorded. A lower percent of hemophilia A carriers who maintain levels of Factor VIII antigen (FVIII:C) >50% at 240 minutes indicates that the laboratory response and sustainment of Factor VIII antigen (FVIII:C) in response to Desmopressin (DDAVP) in adult hemophilia A carriers is reduced as compared to the control group.

SECONDARY OUTCOMES:
Change in the time-course response of Factor VIII antigen levels | Baseline, 240 minutes
  After administration of intravenous Desmopressin (DDAVP) at 0.3mcg/kg, the carriers will be stratified by the type of mutation (mild or severe). The levels of Factor VIII antigen will be measured using a one-stage assay at baseline and 240 minutes. The levels of Factor VIII antigen in hemophilia carriers with mild and severe mutations will be recorded.
Change in the time-course response of von Willebrand factor antigen (vWF:Ag) levels | Baseline, 240 minutes
  After administration of intravenous Desmopressin (DDAVP) at 0.3mcg/kg, the carriers will be stratified by the type of mutation (mild or severe). The levels of von Willebrand factor antigen (vWF:Ag) will be measured using turbidometric assay at baseline and 240 minutes. The levels of von Willebrand factor antigen (vWF:Ag) in hemophilia carriers with mild and severe mutations will be recorded.
Mean FVIII:C/vWF:Ag ratio in subjects with the baseline FVIII:C/vWF:Ag ratio of 1 | 240 minutes
  The sustainment of Factor VIII antigen (FVIII:C) levels in subjects with Factor VIII antigen:von Willebrand factor antigen (FVIII:C:vWF:Ag) ratio of 1will be assessed. The levels of Factor VIII antigen and von Willebrand factor antigen will be measured using a one-stage assay and turbidometric assays respectively. The subjects that have a baseline FVIII:C:vWF:Ag =1 will have their FVIII:C:vWF:Ag ratio assessed at 240 minutes.
Mean FVIII:C/vWF:Ag ratio in subjects with the baseline FVIII:C/vWF:Ag ratio of <1 | 240 minutes
  The sustainment of Factor VIII antigen (FVIII:C) levels in subjects with Factor VIII antigen:von Willebrand factor antigen (FVIII:C:vWF:Ag) ratio of <1 will be assessed. The levels of Factor VIII antigen and von Willebrand factor antigen will be measured using a one-stage assay and turbidometric assays respectively. The subjects that have a baseline FVIII:C:vWF:Ag <1 will have their FVIII:C:vWF:Ag ratio assessed at 240 minutes.
Mean FVIII:C/vWF:Ag ratio in subjects with the baseline FVIII:C/vWF:Ag ratio of >1 | 240 minutes
  The sustainment of Factor VIII antigen (FVIII:C) levels in subjects with Factor VIII antigen:von Willebrand factor antigen (FVIII:C:vWF:Ag) ratio of >1will be assessed. The levels of Factor VIII antigen and von Willebrand factor antigen will be measured using a one-stage assay and turbidometric assays respectively. The subjects that have a baseline FVIII:C:vWF:Ag >1 will have their FVIII:C:vWF:Ag ratio assessed at 240 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sidonio, Jr., MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Hospital of Atlanta Egleston, Atlanta, Georgia
  - Emory University, Atlanta, Georgia